CLINICAL TRIAL: NCT02780947
Title: Prophylactic Substrate Ablation in Post-myocardial Patients Undergoing Defibrillator Implantation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Spyridon Deftereos (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Spyridon Deftereos, Associate Professor of Cardiology, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREVENT-VT study
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure; Myocardial Infarction; Ventricular Tachycardia
Keywords: Ventricular tachycardia; Ablation; Myocardial Infarction; Heart Failure
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic substrate ablation group (Active Comparator): Prophylactic substrate ablation group will undergo substrate mapping and ventricular tachycardia substrate ablation
  Interventions: Procedure: Ventricular tachycardia substrate ablation
- Control group (No Intervention): Control group will undergo substrate mapping

INTERVENTIONS:
Procedure: Ventricular tachycardia substrate ablation — Study protocol
  1. Baseline programmed ventricular stimulation performed from the LV
  2. High density endocardial LV mapping using CARTO® 3 System
  3. Randomized substrate ablation in half patients. Ablation end-point is considered the elimination of all endocardial late and early potentials (LPs and EPs)
  4. Final programmed ventricular stimulation performed from the LV
  Programmed ventricular stimulation with up to 4 extrastimuli from LV is performed and repeated at the end of the procedure in patients undergoing substrate ablation.
  Arms: Prophylactic substrate ablation group

SUMMARY:
Prophylactic substrate ablation in post-MI patients undergoing defibrillator implantation reduces appropriate defibrillator therapies.

DETAILED DESCRIPTION:
Background In patients with Ventricular Tachycardia (VT) and structural heart disease, the Implanted Cardioverter Defibrillator (ICD), provides a significant protection against the risk of sudden death, however it does not prevent arrhythmia recurrences [1-7]. ICD therapies, especially shocks, pose several risks, including decreased quality of life, increased mortality among patients who suffer ICD shock compared with patients who do not and clinically significant anxiety and depression as a result of recurrent ICD shocks, which has been found to occur in more than 50% of patients [8-12]. Furthermore, ICD implantation has been found not to protect against sudden cardiac death in 3-7% of patients [13].

The benefit of novel ICD programming in reducing inappropriate ICD therapy and mortality was demonstrated in Multicenter Automatic Defibrillator Implantation Trial-Reduce Inappropriate Therapy (MADIT-RIT) [14]. Catheter ablation has been considered a plausible curative therapy for VT prevention, especially in patients with VT episodes [15]. The Substrate Mapping and Ablation in Sinus Rhythm to Halt Ventricular Tachycardia (SMASH-VT) and the Ventricular Tachycardia Ablation in Coronary Heart Disease (VTACH) found that prophylactic catheter ablation reduces the incidence of appropriate ICD therapy in patients who had undergone ICD implantation as a means of secondary prevention and had a history of myocardial infarction (MI) [16,17]. It was also shown in a small retrospective study that prophylactic catheter ablation for induced VT reduced the incidence of appropriate ICD therapy in primary prevention post-MI patients [18].

Aim of the study - Statement of Hypothesis Prophylactic substrate ablation in post-MI patients undergoing defibrillator implantation reduces appropriate defibrillator therapies.

ELIGIBILITY:
Inclusion Criteria:

* Post-MI patients eligible for ICD implantation in the setting of primary prevention

Exclusion Criteria:

1. NYHA IV or ambulatory NYHA IV
2. Acute coronary syndrome in the last 40 days
3. Stable angina not eligible to revascularization
4. Revascularization in the last 3 months (except MI)
5. Antiarrhythmic therapy other than b-blockers
6. LVEF<20%
7. GFR<30ml/min/1.73m2
8. Systematic illnesses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Appropriate ICD activation therapies | Within 3 years after ICD implantation
  All post-MI patients will undergo ICD implantation and electroanatomical substrate mapping of the left ventricle. Half patients will also undergo prophylactic VT ablation aiming to late and early potentials elimination.
  Post-MI patients who underwent ICD implantation in the setting of primary prevention and prophylactic substrate ablation will have significant less appropriate ICD therapies.

CONTACTS AND LOCATIONS:
Overall Officials: George Giannopoulos, MD, Principal Investigator — Attikon Hospital, University of Athens; Charis Kossyvakis, MD, Principal Investigator — Athens General Hospital "G. Gennimatas"; Spyros Deftereos, MD, Principal Investigator — Attikon Hospital, University of Athens; Dimitris Tsiachris, MD, Principal Investigator — Athens Heart Center, Athens Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kheiri B, Barbarawi M, Zayed Y, Hicks M, Osman M, Rashdan L, Kyi HH, Bachuwa G, Hassan M, Stecker EC, Nazer B, Bhatt DL. Antiarrhythmic Drugs or Catheter Ablation in the Management of Ventricular Tachyarrhythmias in Patients With Implantable Cardioverter-Defibrillators: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Nov;12(11):e007600. doi: 10.1161/CIRCEP.119.007600. Epub 2019 Nov 8. PMID 31698933